CLINICAL TRIAL: NCT00451048
Title: A Phase II Study of Sunitinib Malate (Sutent®; SU11248) in Patients With Intermediate-2 or High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: Sunitinib in Treating Patients With Myelodysplastic Syndromes or Chronic Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00211; PHL-063 (Other Grant/Funding Number: N01CM62203); CDR0000535656 (Other Grant/Funding Number: N01CM62203); N01CM62203 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-07

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Myelodysplastic Syndromes; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients will receive sunitinib malate (SU11248) by mouth once a day. Treatment may continue for as long as benefit is shown.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with myelodysplastic syndromes or chronic myelomonocytic leukemia. Sunitinib may stop the growth of abnormal cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the overall response rate (complete response, partial response, or hematological improvement) in patients with intermediate-2 or high-risk myelodysplastic syndromes or chronic myelomonocytic leukemia treated with sunitinib malate.

II. Determine the duration of response in patients treated with this drug. III. Determine the overall survival of patients treated with this drug. IV. Determine the progression-free survival of patients treated with this drug. V. Determine the time to disease progression in patients treated with this drug.

VI. Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3-4 weeks and then monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* MDS syndromes meeting 1 of the following: Intermediate-2 disease, high-risk disease (IPSS score>=1.5)
* CMML: WBC>12,000/mm^3, Intermediate-2 disease with WBC=<12,000/mm^3, high-risk disease (IPSS score>=1.5) with WBC=<12,000/mm^3
* Patients with insufficient/inadequate metaphases for cytogenetic analysis are eligible if bone marrow blasts are >10% and/or 2-3 cytopenias are present
* No known brain metastases
* Life expectancy>12 weeks
* ECOG PS 0-2/Karnofsky PS 60-100%
* Calcium=<3.0 mmol/L
* Bilirubin normal
* AST and ALT=<2.5 times upper limit of normal
* Creatinine normal/creatinine clearance>=60 mL/min

Exclusion Criteria:

* No history of significant ECG abnormalities including but not limited to: ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation>=3 beats in a row); QTc prolongation (i.e.QTc interval>=500msec)
* No history of allergic reaction to compounds of similar chemical/biological composition to sunitinib malate
* No NYHA class III-IV congestive heart failure
* Patients with history of NYHA class II congestive heart failure who are asymptomatic on treatment are eligible
* No abdominal fistula/G perforation/intraabdominal abscess within past 28 days
* No serious cardiovascular disease within past 12 months including: cerebrovascular accident or transient ischemic attack, myocardial infarction, cardiac arrhythmia, stable or unstable angina, symptomatic congestive heart failure, coronary or peripheral artery bypass graft or stenting
* No pulmonary embolism within past 12 months
* No uncontrolled hypertension (systolic BP>=140 mmHg/diastolic BP>=90 mmHg)
* No condition impairing ability to swallow/retain sunitinib malate tablets including: GI tract disease resulting in inability to take oral medication, requirement for IV alimentation, prior surgical procedures affecting absorption, active peptic ulcer disease
* No serious/nonhealing wound, ulcer, or bone fracture
* No uncontrolled pre-existing thyroid abnormality
* No concurrent uncontrolled illness including ongoing/active infection
* No psychiatric illness/social situation that would preclude study participation
* Not pregnant/nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* 4 weeks since prior major surgery
* Prior central thoracic radiotherapy that included heart in radiotherapy port allowed provided NYHA congestive heart failure=<class II
* Prior anthracycline exposure allowed provided NYHA congestive heart failure=<class II
* No other prior therapy for MDS/CMML except epoetin alfa, darbepoetin alfa, filgrastim or sargramostim
* At least 2 weeks since prior epoetin alfa
* At least 4 weeks since prior darbepoetin alfa
* No other prior antiangiogenic agents including but not limited to: bevacizumab, sorafenib tosylate, pazopanib hydrochloride, AZD2171, vatalanib, VEGF Trap
* More than 7 days since prior and no concurrent potent CYP3A4 inhibitors
* More than 12 days since prior and no concurrent potent CYP3A4 inducers including: Rifampin, Rifabutin, Carbamazepine, Phenobarbital, Phenytoin, Hypericum perforatum, Efavirenz, Tipranavir
* No concurrent birth control patch/oral birth control pills/depot/injectable birth control methods
* No concurrent therapeutic coumarin-derivative anticoagulants
* Low dose(=<2mg) warfarin for prophylaxis of thrombosis allowed
* Low molecular weight heparin allowed if INR=<1.5
* No concurrent agents with proarrhythmic potential including: Terfenadine, Quinidine, Procainamide, Disopyramide, Sotalol, Probucol, Bepridil, Haloperidol, Risperidone, Indapamide, Flecainide acetate
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2011-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yee, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (4):
- Roswell Park Cancer Institute, Buffalo, New York, United States
- Canada (3):
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients will receive sunitinib by mouth once a day. Treatment may continue for as long as benefit is shown.
  sunitinib malate: Given orally
Period: Overall Study
Arm/Group | Arm I
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 69 [62 to 87]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 1
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response, Partial Response, or Hematologic Improvement) Defined by the International Working Group Criteria
Time Frame: Up to 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 10
percentage of participants | 10

2. Secondary Outcome: Number Participants With Complete, Partial or Hematologic Improvement Response
Description: Assessed by achievement of Complete Response (CR), Partial Response (PR) or Hematologic Improvement (HI)
Time Frame: Up to 6 years
Population: No patient achieved CR, PR or HI as response.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 10
participants | 0

3. Secondary Outcome: Overall Survival
Time Frame: At 6 months and 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 5
months | 13.9 [9.7 to NA] — 95% confidence - 9.7 months to not reached

4. Secondary Outcome: Progression-free Survival
Time Frame: At 6 months and 1 year
Population: Data were not collected
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Progression
Time Frame: At 6 months and 1 year
Population: Date were not collected
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Highest Severity of Observed Adverse Events Assessed by Common Terminology Criteria or Adverse Events Version 3.0 (CTCAE v3.0)
Time Frame: Up to 6 years
Measure: Number; unit: highest grade of adverse event reported
Arm/Group | Arm I
Number analyzed (Participants) | 10
highest grade of adverse event reported | 4

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Encephalitis infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=10)
Anemia (Blood and lymphatic system disorders) | 10
Fatigue (General disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 8
White blood cell decreased (Investigations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less